CLINICAL TRIAL: NCT01375283
Title: Sensory Mapping Following Video-assisted Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kim Wildgaard, MD, Rigshospitalet, Denmark
Other Study IDs: H4-2010-118#2
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Paresthesia; Dysesthesia; Pain
MeSH Terms: conditions — Paresthesia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lung cancer surgery

SUMMARY:
This is a prospective observational cohort study on changes in sensory mapping.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years old
* Elective lung cancer surgery (VATS)

Exclusion Criteria:

* does not understand Danish
* cognitive reduction
* bilateral procedure planned
* previous thoracic surgery
* pregnant or nursing
* known nerve affection from other cause
* alcohol/substance abuse
* inability to cooperate to pain scoring/sensory examination
* > 5 mg methylprednisolone/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing video-assisted thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Area (cm2) | 3 months
  Size of sensory dysfunction

SECONDARY OUTCOMES:
Pain | 3 months
  pain intensity /numerical rating scale)

CONTACTS AND LOCATIONS:
Overall Officials: Mads Werner, MD,, Study Chair — Multidisciplinary Pain Center; Kim Wildgaard, Principal Investigator — Section for Surgical Pathophysiology; Henrik Kehlet, MD, Study Director — Section for Surgical Pathophysiology
Locations (1):
- Section for Surgical Pathophysiology 4074, Copenhagen, Denmark